CLINICAL TRIAL: NCT06849349
Title: INVESTIGATION OF GLYCOPROTEIN, FIBER AND GROWTH FACTOR EXPRESSIONS IN PATIENTS WITH PLACENTA PREVIA, PLACENTA PERFORATA IN THE 3RD TRIMESTER OF PREGNANCY
Brief Title: EXAMINATION OF SOME MOLECULES IN PLACENTAS OF PATIENTS WITH PLACENTA PREVIA, PLACENTA PERCREATA
Status: Recruiting | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: MCBU- Perkreata-previa
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Placenta Percreta, Third Trimester; Placenta Previa
Keywords: Placenta Percreata; Plaenta Previa; GLYCOPROTEIN; FIBER; GROWTH FACTORS
MeSH Terms: conditions — Placenta Accreta; Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 11 Months
Biospecimen Retention: Samples With DNA — placenta tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Pregnant women with Placenta Percreata
- Group 2: Pregnant women with Placenta Previa
- Group 3: Control

SUMMARY:
Placenta previa can cause a risk of severe bleeding during labor. Placenta previa is usually classified into four different types: total, partial, marginal and asymptomatic. The condition is diagnosed by ultrasonography later in pregnancy and its management varies depending on the location of the placenta and the presence of bleeding. Studies show that the increased frequency of placenta previa is associated with increased cesarean section rates and maternal age (1). Furthermore, the effects of placenta previa on maternal and fetal morbidity can be reduced with proper management (2).

Placenta percreata is a condition in which the placenta invades the myometrium (uterine muscle) and serosa (outer surface of the uterus). This can make postpartum detachment of the placenta difficult, leading to severe bleeding and complications. Placenta perforata is often associated with placenta previa and may require surgical intervention. Ultrasonography and magnetic resonance imaging (MRI) are used to diagnose this condition. Risk factors include previous cesarean deliveries and placenta previa (3). Placenta percreata requires careful management as it increases the risk of maternal mortality and morbidity (4).

In this study, we aimed to investigate the levels of decorin, laminin, collagen-1, TGFβ-1, PDGF in placentas of pregnant women with placenta percreata and previa.

DETAILED DESCRIPTION:
In the hospital, blood tests are routinely taken preoperatively from patients hospitalized for placenta percreata and preavia. Blood samples of patients who do not have exclusion criteria and who agree to participate in the study will also be studied from routinely collected blood samples. During the hospitalization of these patients for delivery, following the clamping of the umbilical cord after the birth of the baby (after the bond between the mother and the baby is terminated), 2 ml (one teaspoon) of blood sample will be taken from the cord blood, centrifuged and the serum sample will be separated and stored at -80 degrees. A 3x3 cm piece will be taken from the umbilical cord and placenta (the baby's mate), which will be disposed of as medical waste in the postnatal process, covering all layers. The tissue samples will be placed in a container with 10% formol and preserved. At the time of umbilical cord blood and placenta sampling, these tissues are in a waste state and have no connection with the baby and mother, so there is no harm to the mother or baby during sampling. Tissues (placenta, umbilical cord) and 2 ml (one teaspoon) of blood sample from umbilical cord blood will be taken, centrifuged and serum sample will be separated and stored at -80 degrees Celsius to be used in other similar studies and projects planned to be carried out in the future.

Patients to be selected for the control group will be determined according to the exclusion criteria and will be selected with a similar gestational week and gravida number as the case group (In other studies in the literature, control group patients were collected using this similarity). If the patients selected for the control group give birth at term, tissue samples will be taken. Umbilical cord blood will be collected and stored at -80 and included in the study.

If the patient selected for the control group gives birth prematurely, gives birth in an external center or requests to withdraw from the study, the patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy under 37 weeks
* Age range 18-50
* Being literate in Turkish
* Not having any additional disease
* Agreeing to participate in the study

Exclusion Criteria:

* High-risk pregnancies (gestational hypertension, preeclampsia, HELLP syndrome, chronic hypertension, gestational and pregestational diabetes, cholestasis, intrauterine growth retardation, etc.)

  * Multiple pregnancy
  * Pregnant women under the age of 18
  * Smoking
  * Medication use (excluding routinely used food supplements during pregnancy)
  * Additional disease (thyroid, renal failure, liver failure, hepatitis, heart disease, connective tissue disease, etc.)
  * Immunosuppressive use
  * Presence of active or chronic infection
  * Presence of active or chronic inflammatory disease
  * Patients who gave birth at an external center or later chose to withdraw from the study
  * Patients who did not have any exclusion criteria at the time of Placenta percrata/ placenta previa or when blood was drawn for the control group, but who later developed any exclusion criteria.
  * Premature birth of patients included in the control group

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women of Placenta percreata woman of Placenta previa
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
2% women's with Placenta percreata placenta tissues while birth. Placenta tissues Staining will be Measured by anti-decorin, anti-laminin, anti-collajen-1, anti-TGFβ-1, anti-PDGF immunohistochemistry. | Baseline
maternal and cord blood will be measured TGFB-1 and decorin biochemistry technique. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No